CLINICAL TRIAL: NCT00131495
Title: A Randomized, Double-Blind, Placebo-controlled, Parallel-group, 52-week Study to Evaluate the Efficacy/Safety of Transdermal Patches Delivering Testosterone in Menopausal Women With Low Libido Not Receiving Estrogen Therapy
Brief Title: Study of Transdermal Testosterone Patches in Menopausal Women With Low Libido
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Warner Chilcott (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2004031 and Yr 2 SB
Record Dates: First submitted 2005-08-16; First posted 2005-08-18 (Estimated); Last update posted 2013-04-17 (Estimated); Status verified 2013-04

CONDITIONS: Hypoactive Sexual Desire Disorder
Keywords: Low Libido; Low Desire; Distress
MeSH Terms: conditions — Sexual Dysfunctions, Psychological | interventions — Testosterone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Placebo Comparator): Placebo patch
  Interventions: Drug: Placebo patch
- 2 (Experimental): Testosterone patch (300mcg/day, changed twice a week for one year
  Interventions: Drug: Testosterone (transdermal patches)

INTERVENTIONS:
Drug: Testosterone (transdermal patches) — Testosterone patch (300mcg/day, changed twice a week for one year
  Arms: 2
Drug: Placebo patch — placebo patch changed twice a week for one year
  Arms: 1

SUMMARY:
This study is designed to evaluate the efficacy and safety of 2 doses of the transdermal testosterone patch in naturally or surgically menopausal women with low libido who are not receiving systemic estrogen or estrogen progestin therapy.

DETAILED DESCRIPTION:
Detailed Description:

Hypoactive sexual desire disorder (HSDD) is a condition suffered by as many as 32% of the menopausal population. It is generally defined as a low libido which causes distress. Testosterone therapy (transdermal patch) is currently under investigation for this disorder and results of three phase 3 trials have shown evidence of efficacy in menopausal patients on hormone replacement therapy. Low libido does not discriminate between those women utilizing hormone replacement therapy and those who do not. This study is designed to evaluate the efficacy and safety of 2 doses of the transdermal testosterone patch in naturally or surgically menopausal women with low libido who are not receiving systemic estrogen or estrogen progestin therapy. Persons could elect to go into a single blind study for one year after completing the first yeat double blind

ELIGIBILITY:
Inclusion Criteria:

* Be a generally healthy surgically menopausal woman (12 months), 20 to 70 years of age, not receiving any systemic estrogen or estrogen progestin therapy
* Be a generally healthy naturally menopausal woman (2 years since last period), 40 to 70 years of age, not receiving any systemic estrogen or estrogen progestin therapy.
* Be, in their own judgment, in a stable monogamous sexual relationship for at least one year prior to study entry that is perceived to be secure and communicative with the same partner who is sexually functional and physically present at least 50% of the time.
* Answer affirmatively to ALL of the following questions:

  1. Was the patient's sex life before menopause good and satisfying in general?
  2. Since menopause, has a meaningful loss in the level of desire for sex occurred?
  3. Since menopause, has a significant decrease in sexual activity occurred?
  4. Is the current level of desire for or interest in sex bothering or concerning?
  5. Is an increase in the level of interest in or desire for sex and sexual activity desired?

Exclusion Criteria:

* Physical limitations that would interfere with normal sexual function;
* Estrogen use in the last 12 weeks (vaginal estriol or low dose vaginal estradiol accepted)
* Use of any of the following medications:

  * antiandrogen therapy or topical minoxidil (last 5 years),
  * androgen therapy (past 3 months/implantable past 7 months),
  * systemic corticosteroids,
  * selective serotonin reuptake inhibitors (SSRIs),
  * tricyclic anti-depressants,
  * anti-androgens,
  * systemic beta-blockers,
  * anti-adrenergics,
  * spironolactone,
  * apomorphine,
  * phosphodiesterase type 5 (PDE5) inhibitors (e.g., Viagra, tibolone or selective estrogen receptor modulators (SERMs), including tamoxifen (last 12 weeks))
* Be experiencing any chronic or acute life stress relating to any major life change that may significantly interfere with sexual function;
* Have significant psychiatric disorder (including mild depressive disorder - Beck Depression Inventory-II score of > 14;
* Have current severe dermatological problems or a known suspected hypersensitivity or allergy to any adhesive or any of the constituents of the transdermal testosterone patch
* Have evidence of or history of malignancy (estrogen dependent or any gynecological cancer) within the last 5 years;
* Have diabetes mellitus, active gallbladder disease, unstable thyroid disease, history of cerebrovascular disease, thrombo-embolic disorders, myocardial infarction or angina within the last 5 years or other significant organic disease that would prevent the patient from completing the study, or otherwise affect the outcome of the study.
* Have significant abnormal pretreatment laboratory parameters.

Ages: 20 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 814 (Actual)
Dates: Start 2004-07; Primary Completion 2006-02 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Total satisfying sexual activity over 24 weeks | 6, 12, 24, 36, and 52 weeks

SECONDARY OUTCOMES:
Sexual desire | 6, 12, 24, 36, and 52 weeks
personal distress | 6, 12, 24, 36, and 52 weeks
other domains of the Profile of Female Sexual Function over 24 weeks | 6, 12, 24, 36, and 52 weeks
mood, energy and well-being | 6, 12, 24, 36, and 52 weeks
menopausal symptoms | 6, 12, 24, 36, and 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sue Davis, MD, Principal Investigator — Monash Medical School, The Alfred Hospital
Locations (1):
- Monash Medical School, The Alfred Hospital, Prahran, Victoria, Australia

REFERENCES:
- [Derived] Davis SR, Moreau M, Kroll R, Bouchard C, Panay N, Gass M, Braunstein GD, Hirschberg AL, Rodenberg C, Pack S, Koch H, Moufarege A, Studd J; APHRODITE Study Team. Testosterone for low libido in postmenopausal women not taking estrogen. N Engl J Med. 2008 Nov 6;359(19):2005-17. doi: 10.1056/NEJMoa0707302. PMID 18987368